CLINICAL TRIAL: NCT05729217
Title: Long COVID Symptoms in SARS-CoV-2-positive Children Aged 6-18 Years in China: a Consequential Observation Study
Brief Title: Long COVID Symptoms in SARS-CoV-2-positive Children in China
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tim Shi (Other)
Collaborators: Capital Institute of Pediatrics, China (Other)
Responsible Party: Sponsor-Investigator, Tim Shi, Director, GlobalMD Organization Network Corp
Organization: GlobalMD Organization Network Corp (Other)
Other Study IDs: Children COVID Symptoms
Record Dates: First submitted 2023-02-13; First posted 2023-02-15 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Symptoms and Signs
MeSH Terms: conditions — Signs and Symptoms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1 aged 7-12 years: Group 1 will mainly be primary school students from grade 1 to 6.
  Interventions: Other: SBQ-LC survey
- Group 2 aged 13-15 years: Group 2 will mainly be middle school students from grade 13 to 15.
  Interventions: Other: SBQ-LC survey
- Group 2 aged 16-18 years: Group 3 will mainly be high school students from grade 16 to 18.
  Interventions: Other: SBQ-LC survey

INTERVENTIONS:
Other: SBQ-LC survey — Symptom burden questionnaires of Long COVID

SUMMARY:
The goal of this observational study is to learn about in children aged 6-18 years, after the acute phase of SARS-CoV-2 infection, the COVID symptoms or Long COVID symptoms to impact their daily activities. We aimed to investigate the prevalence of long-lasting symptoms, the duration and intensity of symptoms, quality of life, number of sick days or absences from school, and psychological and social outcomes. The participants will be asked to fill in Long COVID symptom burden questionnaires who had been infected with SARS-CoV-2 as self-reported PRC test or antigen test positive.

DETAILED DESCRIPTION:
The goal of this observational study is to learn about in children aged 6-18 years, after the acute phase of SARS-CoV-2 infection, the COVID symptoms or Long COVID symptoms to impact their daily activities. We aimed to investigate the prevalence of long-lasting symptoms, the duration and intensity of symptoms, quality of life, number of sick days or absences from school, and psychological and social outcomes.

The participants will be asked to fill in SBQ-Long COVID symptom burden survey questionnaires who had been infected with SARS-CoV-2 as self-reported PRC test or antigen test positive.

The survey questionnaires will be filled every two weeks after the participants have been tested SARS-CoV-2 positive.

ELIGIBILITY:
Inclusion Criteria:

infected with SARS-CoV-2 as self-reported PRC test or antigen test positive or have symptoms, but without Covid-19 test.

Exclusion Criteria:

aged below 6 years or above 18 years

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: any children (aged from 6 to 18 years) who had infected with SARS-CoV-2 in Dec. 1st, 2022 to Jan 15th, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
long symptoms of SARS-CoV-2 | 6 to 12 weeks
  the prevalence of long-lasting symptoms, the duration and intensity of symptoms
absences from school | 24 weeks
  number of sick days or absences from school, and psychological and social outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ting Liu, MD, Study Director — Capital Institute of Pediatrics, China; Tim Shi, MD, PhD, Principal Investigator — GlobalMD Organization
Locations (1):
- Capital Institute of Pediatrics, Beijing, China

IPD SHARING:
Plan to Share IPD: No